CLINICAL TRIAL: NCT06406452
Title: A Multi-Center Trial to Assess the Safety and Effectiveness of a Bioresorbable Tracheobronchial Splint in Pediatric Subjects With Clinically Significant Tracheobronchomalacia
Brief Title: Bioresorbable Airway Splint Pivotal Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Materialise (Industry)
Responsible Party: Principal Investigator, Richard Ohye, Professor of Cardiac Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00229974
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tracheobronchomalacia
Keywords: Children; Airway splint; Three-dimensional printed; Multi-stie
MeSH Terms: conditions — Tracheobronchomalacia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bioresorbable Tracheobronchial Splint (Experimental): Participants are admitted to the hospital for this assessment and placement of the splint.
  Interventions: Device: Bioresorbable Tracheobronchial Splint

INTERVENTIONS:
Device: Bioresorbable Tracheobronchial Splint — Subjects will have several imaging and bronchoscopic studies and the placement of the splint will require an open-chest surgery to implant the airway splint (s).
  The Materialise Bioresorbable Tracheobronchial Splint is designed for an individual subject based on Computed Tomography (CT) scans taken using a specific scan protocol. Based on these 3D models, a pre-operative plan is discussed between the Materialise engineering team and the treating surgeon(s) to determine the locations and required dimensions of the splint(s). Each subject may receive up to four splints positioned on subject's trachea or mainstem bronchi.
  Subjects will also have several follow-up visits, and parents will be expected to regularly fill out questionnaires.

SUMMARY:
The purpose of this study is to learn if a three-dimensional (3D) printed airway splint device made to hold open a collapsing airway is a safe and effective treatment of Tracheobronchomalacia (TBM) in children.

The airway splint is bioresorbable, meaning the child's body will absorb the splint over about five years.

DETAILED DESCRIPTION:
Other sites will be added to the registration as sites are on-boarded.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have clinically significant tracheobronchomalacia and:

  1. be unable to wean off of mechanical ventilation, and/or
  2. be currently dependent on a tracheostomy tube, and/or
  3. meet current indications for a tracheostomy or another surgical intervention for TBM
* Subjects must have a life expectancy of at least 2 years, exclusive of TBM
* Subjects must have a parent or legal guardian capable of giving consent on behalf of the subject, and must be willing and able to complete the requirements of clinical trial follow-up
* Subject must have a physician willing to provide follow-up clinical data, including a bronchoscopy at 2 years
* Subjects must be greater than 1 week of age and less than 4 years of age. (Infant subjects born preterm, with low birth weight, or small for gestational age are eligible for trial enrollment if their comorbidities do not present a contraindication to surgical intervention for subjects TBM and airways are of a size that can appropriately be treated with the range of splint sizes offered in this clinical trial)

Patency-Based Pre-Operative Inclusion Criteria:

- Subjects must have tracheobronchomalacia in the trachea, left main bronchus, or right main bronchus a minimum patency of less than 50% in one of these regions

* Screening: In order for a subject to be sent to a clinical trial site for evaluation for the clinical trial, a subject must have tracheobronchomalacia with evidence of less than 50% minimum patency based on a Computed Tomography Scan (CT), Magnetic resonance imaging (MRI), or bronchoscopic exam at referring institution confirmed by an imaging or operative note from the local physician.
* At Enrollment: The subject must have tracheobronchomalacia with minimum patency of less than 50% in the trachea and/or left mainstem bronchus and/or right mainstem bronchus, based on expiration/inspiration CT performed at a clinical trial site performed during visit 1

Intra-Operative Inclusion Criteria:

- The surgeon can safely dissect out the malacic trachea or bronchus/bronchi in order to place the splint

Pre-Operative Exclusion Criteria:

* Subject has significant fixed anatomic tracheal stenosis
* Subject has untreated complete tracheal rings
* Subject has single-lung anatomy
* Subject has single-ventricle cardiac anatomy
* Subject has external compression due to active malignancy, active infection, or an undrained cyst
* Subject has a non-bioresorbable airway stent. Recent removal of any stent will require verification of integrity of the airway wall
* Subject has a contraindication to surgery other than airway compromise
* Subject has a known hypersensitivity to polycaprolactone or hydroxyapatite, and/or a previous unusual reaction to bioresorbable sutures
* Subject has a genetic defect of cartilage formation
* Subject has significant bronchomalacia distal to the mainstem as the predominant source of subject's airway obstruction
* Membranous posterior wall intrusion is the predominant form of collapse

Ages: 1 Week to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects that survive to 6 months post-splinting | 6 months post splint implantation
  All-cause mortality within 6 months (180 days) of splint implantation will count against this endpoint.
The Proportion of splinted regions with equal or greater than (≥) 50% average patency at approximately 4 weeks visit (window ±2 weeks) after splint implantation | Approximately 4 weeks (±2 weeks) post splint implantation
  This will be measured by inspiratory/expiratory cat scan (CT), where average patency is defined as: average cross-sectional area in splinted region on expiration divided by average cross-sectional area in splinted region on inspiration.

SECONDARY OUTCOMES:
The proportion of splinted regions with an absolute increase in average patency of ≥20% from pre-op to approximately 4 weeks visit (window ±2 weeks) post splint implantation | Approximately 4 weeks (±2 weeks) post splint implantation
  This will be measured by inspiratory/expiratory CT, where average patency is defined as: average cross-sectional area in splinted region on expiration divided by average cross-sectional area in splinted region on inspiration.
The proportion of splinted regions with ≥50% minimum patency approximately 4 weeks visit (window ±2 weeks) post splint implantation as measured by video bronchoscopy | Approximately 4 weeks (±2 weeks) post splint implantation
  The percent patency is defined as: observed diameter/expected diameter based upon adjacent non-affected areas x 100, as assessed by the Imaging Core Lab.
The proportion of splinted regions with ≥50% minimum patency 2 years (window ± 4 months) post splint implantation | Approximately 2 years (window ± 4 months) post splint implantation
  The percent patency is defined as: observed diameter/expected diameter based upon adjacent non-affected areas x 100, as assessed by the Imaging Core Lab.
Pediatric Quality of Life Inventory Infant Scales (PedsQL) Pre-operative (pre-op) - up to 1 year visit | Pre-op (prior to splint implementation), up to 1 year visit post splint implantation
  This will be collected for participants (age 0-12 months) This 36-item module measures parent self-reported functioning in physical (6 items), emotional (5 items), social (4 items), and cognitive (5 items) domains, communication (3 items), and worry (5 items), as well as two scales measuring parent-reported family functioning: daily activities (3 items) and family relationships (5 items). Items are reverse-scored and linearly transformed to a 0-100 scale, such that the minimum score is 0 and the maximum score is 100. A higher score indicates better quality of life.
Pediatric Quality of Life Inventory Infant Scales (PedsQL) pre-op - up to 2 year visit | pre-op (prior to splint implementation), up to 2 year visit post splint implantation
  This will be collected for participants (ages 13-24 months). This 45-item module measures parent self-reported physical functioning (9 items), physical symptoms (10 items), emotional functioning (12 items), and social functioning (5 items) domains, cognitive functioning (9 items). Items are reverse-scored and linearly transformed to a 0-100 scale, such that the minimum score is 0 and the maximum score is 100. A higher score indicates better quality of life.
Pediatric Quality of Life Inventory Infant Scales (PedsQL) pre-op - up to 4 year visit | pre-op (prior to splint implementation), up to 4 year visit post splint implantation
  This will be collected for participants (ages 2-4 years). This 21-item module measures parent self-reported physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Items are reverse-scored and linearly transformed to a 0-100 scale, such that the minimum score is 0 and the maximum score is 100. A higher score indicates better quality of life.
Pediatric Quality of Life Inventory Infant Scales (PedsQL) generic core scale post-op 2 year - up to 5 year visit | 2 year, up to 5 year visit post splint implantation
  This will be collected for participants (ages 5-7 years old, 8-12 years) This 23-item module measures parent self-reported physical functioning (8 items), emotional (5 items), social functioning (5 items) and school functioning (5 items). Items are reverse-scored and linearly transformed to a 0-100 scale, such that the minimum score is 0 and the maximum score is 100. A higher score indicates better quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module pre-op | Pre-op (prior to splint implementation)
  There are 36 questions that will be completed from a likert scale of never 0-almost always 4. The Pediatric Quality of Life Family Impact Module (PEDSQL) Score range 0-100. Higher score better quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 3 months post-op | 3 months post splint implantation
  There are 36 questions that will be completed from a likert scale of never 0-almost always 4. The Pediatric Quality of Life Family Impact Module (PEDSQL) Score range 0-100. Higher score better quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 6-months post-op | 6-months post splint implantation
  There are 36 questions that will be completed from a likert scale of never 0-almost always 4. The Pediatric Quality of Life Family Impact Module (PEDSQL) Score range 0-100. Higher score better quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 1 year post-op | 1 year post splint implantation
  There are 36 questions that will be completed from a likert scale of never 0-almost always 4. The Pediatric Quality of Life Family Impact Module (PEDSQL) Score range 0-100. Higher score better quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 2 years post-op | 2 years post splint implantation
  The PedsQL consists of 36 items in eight dimensions: physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 3 years post-op | 3 years post splint implantation
  The PedsQL consists of 36 items in eight dimensions: physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 4 years post-op | 4 years post splint implantation
  The PedsQL consists of 36 items in eight dimensions: physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
Pediatric Quality of Life (PedsQL) Family Impact Module 5 years post-op | 5 years post splint implantation
  The PedsQL consists of 36 items in eight dimensions: physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships that measures health related quality of life. The questionnaire asks how much of a problem each item has been during the past month. Each item is answered on a scale of 0 (never) to 4 (almost always) then the scores are transformed to a 0 to 100 scale, so that higher scores indicate better heath related quality of life.
The proportion of subjects with any device-related complication (DRC) at 6 months' post-implantation. | 6 months post splint implantation
  A DRC will be defined as a subset of Serious Adverse Events (SAE) that are determined to be definitely, probably, or possibly related to the device.
The proportion of subjects with any device-related complication (DRC) at 2 years post splint implantation | 2 years post splint implantation
  A DRC will be defined as a subset of Serious Adverse Events (SAE) that are determined to be definitely, probably, or possibly related to the device

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Ohye, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No